CLINICAL TRIAL: NCT06538636
Title: Prediction Augmented Screening Initiative
Acronym: PASI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: SPLP-001-24S; CX002850 (Other Grant/Funding Number: Veterans Affairs Office of Research & Development)
Record Dates: First submitted 2024-07-30; First posted 2024-08-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Lung Cancer Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The investigators will use a factorial stepped wedge design (SWD) over 15 calendar quarters, with 14 sequence arms and 2 trial sites randomized per sequence to support estimation of separate and combined effects for two intervention types (1-PCP-facing tools and 2-LCS team population management tools). Each half of the arms will sequentially implement one of the interventions, followed by implementation of the second intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Usual Care (No Intervention): Usual care
- PCP facing tools (Experimental): Suite of PCP facing tools activated
  Interventions: Other: PCP-Facing Tools; Other: LCS team population management tools
- LCS team population management tools (Experimental): site-specific dashboard and proactive outreach toolkit
  Interventions: Other: PCP-Facing Tools; Other: LCS team population management tools
- PCP facing tools plus LCS population management dashboard (Experimental): both interventions activated
  Interventions: Other: PCP-Facing Tools; Other: LCS team population management tools

INTERVENTIONS:
Other: PCP-Facing Tools — PCP-facing tools will be turned on as a package: a) enhanced LCS clinical reminder including DP+ generated smart message; b) Integrated one-click DP+ full decision tool for automating personalized information about the net benefit of LCS based on patient characteristics; c) the TurboHM tool: automated Health maintenance app for tracking all preventive care, including a dedicated LCS section with personalized information
  Arms: LCS team population management tools; PCP facing tools; PCP facing tools plus LCS population management dashboard
Other: LCS team population management tools — site-specific dashboard and proactive outreach toolkit
  Arms: LCS team population management tools; PCP facing tools; PCP facing tools plus LCS population management dashboard

SUMMARY:
Lung cancer is responsible for more deaths in the United States than breast, prostate and colon cancer combined and is the number one cancer killer of Veterans. This is because lung cancer is usually diagnosed when the disease has spread, and cure is less likely. Lung cancer screening (LCS) finds cancer at an earlier stage when it is curable, yet only 20% of eligible Veterans have been screened. Uptake is even lower among Black Veterans despite higher lung cancer risk. Using prediction models to identify high-benefit people for whom LCS should be encouraged improves efficiency and reduces disparities. Moreover, it is more patient-centered as shared decision-making conversations can be tailored with personalized information. The US Preventive Services Task Force has called for research to demonstrate that prediction-augmented LCS can be feasibly implemented at the point-of-care. The investigators propose for VA to lead this effort with a large-scale pragmatic clinical trial to show that prediction-augmented LCS is both feasible and improves LCS uptake.

DETAILED DESCRIPTION:
Background: Despite large-randomized trials demonstrating the mortality benefit from lung cancer screening (LCS) and a recommendation from the US Preventive Services Task Force (USPSTF) and VHA since 2013, only 20% of eligible Veterans have received LCS. Uptake is even lower among Black Veterans despite higher lung cancer risk. Current USPSTF eligibility criteria of age and smoking history are simple, but do not incorporate the heterogeneity in lung cancer risk and life expectancy across people and leads to exclusion of some persons, especially Blacks, with potential for high benefit from LCS. While the USPSTF acknowledged that using prediction models to augment simple eligibility criteria is more efficient and equitable, they stopped short of recommending prediction-augmented LCS, noting that a pragmatic trial was needed to demonstrate that prediction-augmented LCS can be feasibly implemented in real-world settings and assess its impact on LCS uptake. Significance: By demonstrating the real-world feasibility of prediction-augmented LCS, and its ability to improve LCS uptake especially in those of high-benefit, the VA as a learning healthcare system will influence national LCS guidelines and improve LCS outcomes both inside and outside the VA. Innovation & Impact: Prediction-augmented LCS is based on strong evidence, yet implementing this approach would represent paradigm shift from typical preventive cancer screening. The proposed work is a unique opportunity for the VA to advance implementation of more equitable, personalized LCS by improving on the status quo of making broad 'one-size-fits-all' recommendations. The innovation is the advancement of primary care-facing and population management informatics tools that present individualized information on how strongly to encourage LCS, with the potential to be expanded to other cancer screenings. Specific Aims: 1. Conduct a pragmatic stepped wedge (site-level) factorial trial comparing usual care (USPSTF criteria) versus prediction-augmented LCS (supported by primary care-facing informatics tools, LCS team population management tools, external facilitation) on effectiveness at increasing LCS uptake. 2. Determine what drives implementation success of prediction-augmented LCS in various contexts, using mixed methods. Methodology: The investigators will utilize a factorial stepped wedge design in the Lung Precision Oncology Program network to establish the effectiveness and evaluate the implementation of precision-augmented LCS. Veterans assigned a PCP at a participating site and who meet inclusion criteria based on Clinical Data Warehouse data will be passively enrolled in the study: 1) patients meeting USPSTF criteria for LCS; OR 2) patients whose predicted LCS benefit exceeds a stringent high-benefit threshold of life gained with annual LCS (to capture high-benefit Veterans currently excluded by USPSTF criteria). The primary outcome is the percentage of eligible subjects who complete LCS during each study quarter. The factorial design allows us to discern the effect on LCS uptake of primary care-facing vs LCS team population management tools. Secondary outcomes include uptake among Veterans with the highest predicted benefit from LCS, uptake among high-benefit Black Veterans, effects on lung cancer detection rates, LCS outcomes (e.g., invasive procedures, complications) and projected lung cancer deaths avoided among additional people screened due to the interventions, and care gaps in which LCS was ordered but not completed. Implementation evaluation will be guided by the i-PARIHS framework using mixed methods. This approach combines data drawn from across all trial sites (tool usage data, clinician surveys, facilitation data, patient interviews) to gain a broad view of implementation, with in-depth ethnographic assessments from 6 selected sites that will provide deeper insights into how and why implementation succeeded (or faced challenges) in different contexts. Our findings will inform creation of an implementation playbook to support enterprise-wide spread of prediction-augmented LCS. Next Steps / Implementation: The investigators will work with our operational partners to spread implementation of prediction-augmented LCS across the VA enterprise.

ELIGIBILITY:
Inclusion Criteria:

Veterans assigned a PCP at a participating site and who meet inclusion criteria at any point during the study timeframe will be enrolled into the trial. There will be two paths to patient inclusion:

* meeting USPSTF eligibility criteria for LCS, as currently encoded in the background logic of LCS clinical reminders maintained by the VA National Center for Lung Cancer Screening (i.e., age 50-80 years; smoked 20 pack-years; current smoking or quit <15 years ago) OR
* predicted benefit calculated using LYFS-CTVA model exceeds a stringent high-benefit threshold of life-year gains with annual LCS, as recommended in the 2021 CHEST LCS guidelines

Exclusion Criteria:

* Veterans who have previously undergone lung cancer screening, are diagnosed with lung cancer, or who do not meet eligibility criteria outlined above

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23520 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-05 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
LDCT receipt | From time of intervention activation at the facility to the receipt of LDCT scan up to 169 weeks
  the probability of receiving an initial LDCT LCS scan at a given site among eligible subjects during each quarter of the study (quarter assigned by date of the LDCT order as this event is most proximal to the LCS decision; passage of time between order and scan completion could lead to erroneous attribution of primary outcome to the wrong study phase if scan date is used

SECONDARY OUTCOMES:
High-benefit Veteran Uptake | Every quarterly through study completion, an average of 3 years
  LCS orders and uptake among high-benefit Veterans
Black Veteran Uptake | Every quarterly through study completion, an average of 3 years
  LCS orders and uptake among high-benefit Black Veterans
non-high-benefit uptake | Every quarterly through study completion, an average of 3 years
  LCS orders and uptake among eligible but non-high-benefit Veterans and among those with high comorbidity
Lung cancer detection | Every quarterly through study completion, an average of 3 years
  lung cancer detection rates
Invasive procedures | Every quarterly through study completion, an average of 3 years
  invasive procedures resulting from lung cancer screening exam findings
Complications from invasive procedures | quarterly through study completion, an average of 3 years
  Complications following invasive procedures done as a result of LCS
lung cancer deaths avoided | through study completion, an average of 3 years
  this will be calculated among additional people screened due to study interventions

CONTACTS AND LOCATIONS:
Overall Officials: Nichole T Tanner, MD MS BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (4):
- United States (4):
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No